CLINICAL TRIAL: NCT01652911
Title: A Phase I/II Study of the Safety and Efficacy of Sernova's Cell PouchTM for Therapeutic Islet Transplantation
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Sernova Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00028097
Record Dates: First submitted 2012-07-12; First posted 2012-07-30 (Estimated); Last update posted 2022-05-11 (Actual); Status verified 2016-07

CONDITIONS: Type I Diabetes
Keywords: Islet Transplantation; Cell Pouch
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cell Pouch (Experimental): Participants with Type-1 diabetes will receive the Sernova Cell Pouch™ implanted in the subcutaneous site, two to approximately twelve weeks prior to transplantation of islets into the Cell Pouch™.
  Interventions: Device: Sernova Cell Pouch

INTERVENTIONS:
Device: Sernova Cell Pouch — The Cell Pouch™ is an implantable medical device for transplantation of donor islets for Type-1 diabetes as an alternative to the current standard of care using intraportal delivery of islets.

SUMMARY:
This is an open-label, single arm, non-randomized safety and efficacy study, where participants with Type-1 diabetes will receive the Sernova Cell Pouch™ implanted in the subcutaneous site, two to approximately twelve weeks prior to transplantation of islets into the Cell Pouch™.

The primary objective of this study is to assess the safety of the Sernova Cell Pouch™ in adult participants with Type-1 diabetes receiving islet transplantation for the first time.

Secondary objectives are the following:

1. To determine the proportion of subjects implanted with the Cell Pouch™ and transplanted with islets into the Cell Pouch™ who achieve and maintain insulin independence after islet transplantation.
2. To obtain preliminary data on the efficacy of the Cell Pouch™ to maintain adequate immunological protection against both allo- and autoimmunity of islet transplant recipients.
3. To determine through retrospective analysis comparative metabolic function and engraftment efficiency using patients undergoing standard intraportal islet transplantation under the current alemtuzumab standard of care protocol.

ELIGIBILITY:
Inclusion Criteria:

To be eligible the participant must have had T1DM for more than 5 years, complicated by at least 1 of the following situations that persist despite intensive insulin management efforts:

1. Reduced awareness of hypoglycemia, as defined by the absence of adequate autonomic symptoms at plasma glucose levels < 3.0 mmol/L, indicated by, 2 or more episodes of severe hypoglycemia requiring third party assistance within 12 months, a Clarke score ≥4, HYPO score ≥1,000, lability index (LI) ≥400 or combined Hypo/LI >400/300
2. Metabolic instability, characterized by erratic blood glucose levels that interfere with daily activities and or 2 or more hospital visits for diabetic ketoacidosis over the last 12 months.

Participants must be capable of understanding the purpose and risks of the study and must sign a statement of informed consent.

Exclusion Criteria:

1. Severe co-existing cardiac disease, characterized by any one of these conditions: (a) recent myocardial infarction (within past 6 months); (b) left ventricular ejection fraction <30%; or (c) evidence of ischemia on functional cardiac exam.
2. Active alcohol or substance abuse, to include cigarette smoking (must be abstinent for 6 months prior to transplant).
3. Psychiatric disorder making the subject not a suitable candidate for transplantation, (e.g., schizophrenia, bipolar disorder, or major depression that is unstable or uncontrolled on current medication).
4. History of non-adherence to prescribed regimens.
5. Active infection including Hepatitis C, Hepatitis B, HIV, TB (subjects with a positive PPD performed within one year of enrollment, and no history of adequate chemoprophylaxis).
6. Any history of or current malignancies except squamous or basal skin cancer.
7. BMI > 35 kg/m2 at screening visit.
8. Age less than 18 or greater than 68 years.
9. Measured glomerular filtration rate (GFR) <60 mL/min/1.73 m2.
10. Presence or history of macroalbuminuria (>300 mg/g creatinine).
11. Clinical suspicion of nephritic (hematuria, active urinary sediment) or rapidly progressing renal impairment (e.g. Increase in serum creatinine of 25% within the last 3-6 months).
12. Baseline Hb < 105g/L in women, or < 120 g/L in men.
13. Baseline screening liver function tests outside of normal range, with the exception of uncomplicated Gilbert's Syndrome. An initial LFT panel with any values >1.5 times the upper limit of normal (ULN) will exclude a patient without a re-test; a re test for any values between ULN and 1.5 times ULN should be made, and if the values remain elevated above normal limits, the patient will be excluded.
14. Untreated proliferative retinopathy.
15. Positive pregnancy test, intent for future pregnancy or male subjects' intent to procreate, failure to follow effective contraceptive measures, or presently breast feeding.
16. Previous transplant or evidence of significant sensitization on PRA (at the discretion of the investigator).
17. Insulin requirement >1.0 U/kg/day
18. HbA1C >12%.
19. Uncontrolled hyperlipidemia [fasting LDL cholesterol > 3.4 mmol/L, treated or untreated; and/or fasting triglycerides > 2.3 mmol/L].
20. Under treatment for a medical condition requiring chronic use of steroids.
21. Use of coumadin or other anticoagulant therapy (except aspirin) or subject with PT INR > 1.5.
22. Untreated Celiac disease.
23. Patients with Graves disease will be excluded unless previously adequately treated with radioiodine ablative therapy.
24. Any medical condition that, in the opinion of the clinical investigator, will interfere with the safe participation in the trial.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
To assess the safety of the Sernova Cell Pouch™ in adult participants with Type-1 diabetes receiving islet transplantation for the first time. | 3 years post-initial Cell Pouch™ implant.
  A tracking log will document adverse events with grading classification as per protocol. For the primary objective endpoint, safety will be assessed following initial Cell Pouch implantation, at the time of islet transplantation, and approximately one month following the initial islet transplantation. Safety will further be assessed at approximately three, six, nine and twelve months and then yearly thereafter.

SECONDARY OUTCOMES:
To determine the proportion of subjects implanted with the Cell Pouch™ and transplanted with islets into the Cell Pouch™ who achieve insulin independence after islet transplantation. | 3 years post-initial Cell Pouch™ implant.
  The proportion of study participants achieving and maintaining insulin independence (c-peptide, HbA1c level) with good glycemic control (blood sugar measurement) at 1, 3, 6 and 12 months and yearly thereafter.
To obtain preliminary data on the efficacy of the Cell Pouch™. | 3 years post-initial CellPouch™
  The efficacy analysis will compare observed proportion of subjects who become insulin independent at the end of month 3 following the completed islet transplant. The outcomes will also be analyzed at 1, 6 and 12 months and then yearly thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: James Shapiro, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta - Clinical Islet Transplant Program, Edmonton, Alberta, Canada

REFERENCES:
- See also: Related Info — http://www.islet.ca
- See also: Related Info — http://www.sernova.com